CLINICAL TRIAL: NCT00002579
Title: PROTOCOL FOR THE SCOTTISH CHEMO-ENDOCRINE TRIAL D
Brief Title: Tamoxifen Following Combination Chemotherapy in Treating Women With Operable Invasive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scottish Cancer Therapy Network (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063694; SCTN-BR9403; EU-94004
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Fluorouracil; Methotrexate; Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: fluorouracil
Drug: methotrexate
Drug: tamoxifen citrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Combining combination chemotherapy with hormone therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without tamoxifen in treating women with stage I or stage II breast cancer that can be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the disease-free and overall survival produced by adjuvant tamoxifen given after postoperative chemotherapy with cyclophosphamide/methotrexate/fluorouracil (CMF) vs. adjuvant CMF alone in women with primary breast cancer.

OUTLINE: This is a randomized study. Patients are stratified by age and by participating institution. All patients undergo surgical resection with local radiation therapy, as appropriate. Within 4 weeks of surgery, patients receive cyclophosphamide, methotrexate, and fluorouracil (CMF) every 3 weeks for 6 courses. Radiotherapy is given within 4 weeks of completion of CMF. Before beginning the last course of CMF, patients are randomized to receive either oral tamoxifen daily for 5 years or no further therapy. Patients are followed every 6 months for 5 years, then yearly. Hormone therapy is prohibited except as specified above and except for short-term hormone replacement therapy for severe unresponsive menopausal symptoms.

PROJECTED ACCRUAL: Approximately 2,000 patients will be required. Data on patients entered in Scotland as part of this study will be pooled with data from the EORTC-10901 study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed breast cancer with palpable, unilateral, invasive disease Bilateral mammography required within 1 year prior to randomization TNM Stage T1-3, N0-1, M0 disease for which adjuvant chemotherapy is considered an essential part of initial therapy No prior pure in situ carcinoma in either breast No concurrent in situ carcinoma only No Paget's disease of the nipple without underlying invasion No evidence of distant disease, e.g.: No ipsilateral supraclavicular node enlargement unless proven benign Hormone receptor status: Any status

PATIENT CHARACTERISTICS: Age: Not specified Sex: Women only Menopausal status: Pre- or postmenopausal Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No serious unrelated illness No prior invasive malignancy at any other site except adequately treated nonmelanomatous skin cancer No pregnant or nursing women Adequate contraception required

PRIOR CONCURRENT THERAPY: No prior tamoxifen and not currently receiving tamoxifen

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 1993-03

CONTACTS AND LOCATIONS:
Overall Officials: W.D. George, MD, MS, FRCS, Study Chair — University of Glasgow
Locations (10):
- United Kingdom (10):
  - Leicester Royal Infirmary NHS Trust, Leicester, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - University of Glasgow, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Ayr Hospital, Ayr
  - Falkirk Royal Infirmary, Falkirk